CLINICAL TRIAL: NCT07363590
Title: A Dose Escalation Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-1045 in Participants With Systemic Lupus Erythematosus and Rheumatoid Arthritis
Brief Title: A Clinical Study of MK-1045 in People With Lupus or Rheumatoid Arthritis (MK-1045-004)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1045-004; U1111-1326-4816 (Registry Identifier: UTN); 2025-523412-36-00 (Registry Identifier: EU CT); MK-1045-004 (Other: MSD)
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 Prime Dose Escalation Panels (Experimental): Participants will receive single intravenous (IV) doses of MK-1045 at varying dose levels.
  Interventions: Biological: MK-1045
- Part 2 Step-up Dose Escalation Panels (Experimental): Participants will receive 3 step up doses of MK-1045 as a prime, step-up and target dose over a 3-week dosing interval.
  Interventions: Biological: MK-1045
- Part 3 Dose Expansion Panels (Optional) (Experimental): Participants will receive 3 step up doses of MK-1045 as a prime, step-up and target dose over a 3-week dosing interval.
  Interventions: Biological: MK-1045

INTERVENTIONS:
Biological: MK-1045 — IV infusion
  Other Names: CN201

SUMMARY:
This study looks at a study medicine called MK-1045 in people with lupus and rheumatoid arthritis (RA). The main goal of the study is to learn about the safety of MK-1045 and if people tolerate it when they receive it at different dose levels (amounts).

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index between 18 and 32 kg/m^2, inclusive
* Systemic lupus erythematosus (SLE): Has a diagnosis of SLE for at least 6 months and met the European Alliance of Associations for Rheumatology (EULAR)/ American College of Rheumatology (ACR) 2019 classification criteria
* SLE: Is taking at least one background therapy for SLE
* RA: Has a diagnosis of RA for at least 6 months and meets the 2010 ACR-EULAR classification criteria for RA

Exclusion Criteria:

* Has a known active infection (excluding fungal infection of nail beds), or any major episode of infection requiring hospitalization or treatment with anti-infectives within 8 weeks prior to the Day 1 dosing
* History of serious recurrent or chronic infection
* Is known to be infected with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus
* Has evidence of active tuberculosis (TB), latent TB, or inadequately treated TB
* Has a significant or uncontrolled medical disease in any organ system not related to RA or SLE
* For RA participants, has a history of any arthritis with onset before age 17 years
* Has a current inflammatory condition other than SLE or RA that could interfere with disease activity assessments
* History of cancer (except fully treated nonmelanoma skin cancers or cervical carcinoma in situ after complete surgical removal) and is disease free for <5 years before Day 1 dosing
* Has had a major surgery within 3 months prior to Screening or has a major surgery planned during the study.
* Has symptomatic heart failure (New York Heart Association class III or IV) or myocardial infarction or unstable angina pectoris within 6 months prior to Screening
* Has a severe chronic pulmonary disease requiring oxygen therapy
* Has current active lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-07-16 (Estimated); Study Completion 2029-07-16 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with One or More Adverse Events (AEs) | Up to approximately 12 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Part 1: Number of Participants who Discontinue Study Drug Due to an AE | Up to approximately 4 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Part 2 and Part 3: Number of Participants with One or More AEs | Up to approximately 52 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Part 2 and Part 3: Number of Participants who Discontinue Study Drug Due to an AE | Up to approximately 2 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

SECONDARY OUTCOMES:
Part 1: Maximum Serum Concentration (Cmax) of MK-1045 | At designated time points up to 12 weeks
  Blood samples will be collected to determine the Cmax, obtained directly from the measured value of the plasma concentration-time curve.
Part 1: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-1045 | At designated time points up to 12 weeks
  Blood samples will be collected to determine the AUC0-Inf of MK-1045.
Part 1: Percentage of Participants with a Peripheral B Cell Count Less Than the Lower Limit of Quantitation (LLOQ) at the End of Each Treatment Period | At designated time points up to 12 weeks
  Blood samples will be collected to determine the B cell depletion in peripheral blood after treatment with MK-1045.
Part 2 and Part 3: Cmax of MK-1045 | At designated time points up to 52 weeks
  Blood samples will be collected to determine the Cmax, obtained directly from the measured value of the plasma concentration-time curve.
Part 2 and Part 3: Area Under the Concentration-Time Curve From Time 0 to the End of the Dosing Interval (AUCtau) of MK-1045 | At designated time points up to 52 weeks
  Blood samples will be collected to determine the AUCtau of MK-1045.
Part 2 and Part 3: Percentage of Participants with a Peripheral B Cell Count Less Than the LLOQ at the End of the Treatment Period | At designated time points up to 52 weeks
  Blood samples will be collected to determine the B cell depletion in peripheral blood after treatment with MK-1045.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com